CLINICAL TRIAL: NCT00592098
Title: A Double-Blind, Placebo-Controlled Cross-Over Study to Evaluate the Efficacy of 2PX (Topical Strontium Chloride Hexahydrate) in Patients With Persistent, Moderate-to-Severe Lower Limb Post-Amputation Stump Pain.
Brief Title: 2PX (Topical Strontium Chloride Hexahydrate) in Patients With Post-Amputation Stump Pain.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SantoSolve AS (Industry)
Responsible Party: Thorfinn Ege, SantoSolve AS
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMR-1589 / 2PX-SP-01; EUDRACT no: 2006-005447-29
Record Dates: First submitted 2007-12-29; First posted 2008-01-11 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2007-12

CONDITIONS: Amputation Stumps; Pain
Keywords: Lower limb amputation at least 6 months prior to inclusion; Presenting with moderate-to-severe pain intensity; Outpatients, aged 18 years and above
MeSH Terms: conditions — Pain | interventions — strontium chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 2PX
  Interventions: Drug: Strontium chloride hexahydrate
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Strontium chloride hexahydrate — Cutaneous solution, 1 ml dose per 100 sq cm of affected skin area, To be applied twice daily for 28 days.
  Other Names: 2PX
  Arms: 1
Drug: Placebo — Cutaneous saline solution, 1 ml dose per 100 sq cm of affected skin area, To be applied twice daily for 28 days.
  Arms: 2

SUMMARY:
The objective of this study is to investigate the analgesic effect of topical strontium chloride in stump pain, and to prospectively determine other efficacy and safety measures of topical strontium chloride in stump pain.

ELIGIBILITY:
Inclusion Criteria:

* Lower limb amputation at least 6 months prior to inclusion
* Presenting with moderate-to-severe pain intensity (above 50 on 100 mm VAS) at screening, to be confirmed prior to randomisation as: Mean (over the 14 days run-in period) stump API rating above 50 on a 100 mm VAS
* Outpatients, aged 18 years and above
* Written informed consent

Exclusion Criteria:

* Subjects who have received treatment with any potent opioid in the 4 weeks prior to study entry (i.e. an opioid assumed to cause abstinence symptoms upon abrupt cessation)
* Subjects taking any analgesic medication (except for rescue medication as defined in this protocol)
* Subjects with expressed dissatisfaction with their prosthesis comfort
* Pregnant or breast-feeding women
* Any malignant disease
* Subjects who have received an investigational drug or used an investigational device in the 30 days prior to study entry.
* Subjects unable to comply with the study assessments
* Subjects with documented or suspected alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Average Pain Intensity (API): will be measured each evening in response to the question: 'What was your average pain intensity over the past 24 hours?' on a 100 mm VAS (0 = no pain, 100 = worst pain imaginable). | 24 hours

SECONDARY OUTCOMES:
• Worst Pain Intensity (WPI) | 24 hours
• Pain relief | Weekly
• Sleep disturbance | 24 hours
• Use of rescue medication | Daily
• Patient Global Impression of Change (PGIC) | Weekly
• Prosthesis bothersomeness | Weekly
• Quality of life assessment | Q 14 days
Local skin irritability | Q 14 days
Adverse events | Q 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Knut T Smerud, MSc, Study Director — Smerud Medical Research International AS, Drammensveien 41, N-0271 Oslo, Norway
Locations (1):
- Smerud Investigator site 1, Oslo, Norway